CLINICAL TRIAL: NCT02970669
Title: Multicenter, Randomized, Double-blind, Double Dummy, Parallel Group, Active-controlled 8-week Study and 8-week Open Label Extension to Evaluate the Effect of Initiation of Sacubitril/Valsartan on Objective Measures of Waking Activity and Sleep, as Health-related Quality of Life Functions in Subjects With Heart Failure and Reduced Ejection Fraction (AWAKE-HF).
Brief Title: Study on the Effects of Sacubitril/Valsartan on Physical Activity and Sleep in Heart Failure With Reduced Ejection Fraction Patients.
Acronym: AWAKE-HF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CLCZ696BUS14
Expanded Access: NCT02389933 (No longer available)
Record Dates: First submitted 2016-11-17; First posted 2016-11-22 (Estimated); Results first posted 2019-04-08 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2021-10

CONDITIONS: Heart Failure, Reduced Ejection Fraction
Keywords: Heart failure with reduced left ventricular ejection fraction (LVEF); Cardiac dysfunction; Heart muscle dysfunction; Left ventricular (LV) dilation; Left ventricular hypertrophy; HF; AHF; CHF; acute heart failure; chronic heart failure; congestive heart failure; congestive cardiac failure; Heart failure; HReEF; Physical Activity; Actigraphy; Home sleep test; wake
MeSH Terms: conditions — Heart Failure, Systolic; Dilatation, Pathologic; Hypertrophy, Left Ventricular; Heart Failure; Motor Activity | interventions — sacubitril; Valsartan; sacubitril and valsartan sodium hydrate drug combination; Enalapril

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Enalapril (Active Comparator): Double blind treatment epoch: Patients randomized to this arm received 1 tablet of enalapril and 1 tablet of matching placebo sacubitril/valsartan twice daily for 8 weeks. All Patients began the study on Dose Level 1 (i.e. 2.5 mg enalapril BID). Patients may have been sequentially up-titrated to achieve desired dose of Dose Level 3 (i.e. 10 mg enalapril BID). Patients not tolerating dose escalation could have been titrated down to next lower dose level.
  Open-label treatment epoch: All patients entering this epoch (8 weeks) were given sacubitril/valsartan 49/51 mg BID (Dose Level 2) unless they completed the double-blind treatment epoch on enalapril Dose Level 1. Instead, these patients entered open-label epoch on Dose Level 1 of sacubitril/valsartan. Patients may have been sequentially up-titrated to achieve desired dose of Dose Level 3 of sacubitril/valsartan. Patients not tolerating dose escalation could have been titrated down to next lower dose level.
  Interventions: Drug: sacubitril/valsartan (LCZ696); Drug: enalapril; Drug: matching placebo sacubitril/valsartan (LCZ696)
- Sacubitril/Valsartan (Experimental): Double blind treatment epoch: Patients randomized to this arm received 1 tablet of sacubitril/valsartan and 1 tablet of matching placebo enalapril twice daily for 8 weeks. All Patients began the study on Dose Level 1 (i.e. 24/26 mg sacubitril/valsartan BID). Patients may have sequentially been up-titrated to achieve desired dose of Dose Level 3 (i.e. 97/103 mg sacubitril/valsartan BID). Patients not tolerating dose escalation could have been titrated down to next lower dose level.
  Open-label treatment epoch: All patients entering this epoch (8 weeks) were given sacubitril/valsartan 49/51 mg BID (Dose Level 2) unless they completed the double-blind treatment epoch on Dose Level 1. Instead, these patients entered open-label epoch on Dose Level 1. Patients may sequentially have been up-titrated to achieve desired dose of Dose Level 3. Patients not tolerating dose escalation could have been titrated down to next lower dose level.
  Interventions: Drug: sacubitril/valsartan (LCZ696); Drug: matching placebo enalapril

INTERVENTIONS:
Drug: sacubitril/valsartan (LCZ696) — sacubitril/valsartan tablet taken orally.
Drug: enalapril — Enalapril tablet taken orally.
  Arms: Enalapril
Drug: matching placebo sacubitril/valsartan (LCZ696) — matching placebo sacubitril/valsartan tablet taken orally
  Arms: Enalapril
Drug: matching placebo enalapril — matching placebo enalapril tablet taken orally
  Arms: Sacubitril/Valsartan

SUMMARY:
The purpose of this study was to investigate the effects of initiation of sacubitril/valsartan vs enalapril treatment on objective measures of both waking activity and sleep in subjects with heart failure with reduced ejection fraction.

ELIGIBILITY:
Key Inclusion Criteria:

* Written informed consent must be obtained before any assessment is performed.
* Men and women between 18 and 80 years of age
* Subjects diagnosed with NYHA class II or III heart failure and with reduced ejection (HFrEF).

(Reduced ejection is defined as left ventricular EF ≤ 40%. LVEF ≤40% may be determined via any local measurement within the past 6 months prior to signing consent, using echocardiography, multi gated acquisition scan (MUGA), CT scanning, MRI or ventricular angiography provided no subsequent study documenting an EF of >40%. If the EF measurement is expressed as a value range, the average of the range endpoint values should be used as the EF).

* Subjects must be a candidate for treatment with sacubitril/valsartan as per USPI.
* Subjects must be living in a traditional residence, apartment, or non-communal adult home where they can move about freely and frequently and are primarily responsible for scheduling their sleep and daily activities.

Key Exclusion Criteria:

* Subjects with a history of hypersensitivity to any of the study drugs, including history of hypersensitivity to drugs of similar chemical classes, or allergy to ACEIs, ARBs, or NEP inhibitors as well as known or suspected contraindications to the study drugs.
* Subjects with a history of angioedema drug related or otherwise
* Subjects with symptomatic hypotension or systolic blood pressure <100 mmHg at screening or <95 mmHg at randomization
* Subjects with any conditions in skin or upper extremities which would limit the ability to tolerate a wrist-worn actigraphy device on the non-dominant arm for 24 hours/day for the duration of the study.
* Subjects who are non-ambulatory or use mobility assistive devices such as motorized devices, wheelchairs, or walkers. The use of canes for stability while ambulating is acceptable.
* Subjects with physical activity impairment primarily due to conditions other than heart failure such as:
* Exertional angina inflammatory or degenerative joint disease -gout
* peripheral vascular disease
* neurologic disease affecting activity or mobility

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2016-12-16 (Actual); Primary Completion 2018-03-19 (Actual); Study Completion 2018-03-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (23):
- United States (23):
  - Novartis Investigative Site, Fort Payne, Alabama
  - Novartis Investigative Site, Beverly Hills, California
  - Novartis Investigative Site, Stockton, California
  - Novartis Investigative Site, West Hills, California
  - Novartis Investigative Site, Doral, Florida
  - Novartis Investigative Site, Inverness, Florida
  - Novartis Investigative Site, Ormond Beach, Florida
  - Novartis Investigative Site, Port Orange, Florida
  - Novartis Investigative Site, Lutherville, Maryland
  - Novartis Investigative Site, East Brunswick, New Jersey
  - Novartis Investigative Site, Ridgewood, New Jersey
  - Novartis Investigative Site, Columbia, South Carolina
  - Novartis Investigative Site, Greenville, South Carolina
  - Novartis Investigative Site, Lancaster, South Carolina
  - Novartis Investigative Site, Allen, Texas
  - Novartis Investigative Site, McKinney, Texas
  - Novartis Investigative Site, New Braunfels, Texas
  - Novartis Investigative Site, San Antonio, Texas
  - Novartis Investigative Site, San Marcos, Texas
  - Novartis Investigative Site, Sherman, Texas
  - Novartis Investigative Site, Tomball, Texas
  - Novartis Investigative Site, Midlothian, Virginia
  - Novartis Investigative Site, Tacoma, Washington

REFERENCES:
- [Derived] Khandwalla RM, Grant D, Birkeland K, Heywood JT, Fombu E, Owens RL, Steinhubl SR; AWAKE-H. F. Study Investigators. The AWAKE-HF Study: Sacubitril/Valsartan Impact on Daily Physical Activity and Sleep in Heart Failure. Am J Cardiovasc Drugs. 2021 Mar;21(2):241-254. doi: 10.1007/s40256-020-00440-y. Epub 2020 Sep 26. PMID 32978755
- See also: A Plain Language Trial Summary is available on novartisclinicaltrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=471

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 140 subjects from 23 sites in the US were randomized. The study consisted of a 2-week baseline period , followed by an 8-week double-blind treatment period ( randomized to sacubitril/valsartan or enalapril, in a 1:1 ratio), followed by an 8-week open label extension period during which all patients were treated with sacubitril/valsartan.
Period: Double-blind Period
Arm/Group | Enalapril | Sacubitril/Valsartan
Started (Randomized) | 70 | 70
Completed | 62 | 64
Not Completed | 8 | 6
Not completed — Adverse Event | 4 | 0
Not completed — Death | 1 | 0
Not completed — Study terminated by sponsor | 1 | 2
Not completed — Physician Decision | 0 | 2
Not completed — Withdrawal by Subject | 2 | 2
Period: Open-label Period
Arm/Group | Enalapril | Sacubitril/Valsartan
Started | 62 | 64
Completed | 58 | 62
Not Completed | 4 | 2
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Adverse Event | 1 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Enalapril: Double-blind Treatment Period (Week 1 - Week 8): Enalapril Open-label Treatment Period (Week 9 - Week 16): Sacubitril/Valsartan
- Sacubitril/Valsartan: Double-blind Treatment Period (Week 1 - Week 8): Sacubitril/Valsartan Open-label Treatment Period (Week 9 - Week 16): Sacubitril/Valsartan
- Total: Total of all reporting groups
Arm/Group | Enalapril | Sacubitril/Valsartan | Total
Number analyzed (Participants) | 70 | 70 | 140
Age, Continuous [Mean (Full Range); unit: years] | 64.2 [26 to 81] | 62.3 [45 to 80] | 63.3 [26 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 18 | 32
  Male | 56 | 52 | 108
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 60 | 48 | 108
  Black | 8 | 13 | 21
  Asian | 1 | 4 | 5
  Native American | 0 | 1 | 1
  Pacific Islander | 0 | 1 | 1
  Other | 1 | 2 | 3
  Unknown | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Ratio of Mean Activity Counts Collected During the Most Active 30 Minutes of the Subject's Day Between Week 8 and Baseline
Description: The primary endpoint is the ratio in mean activity counts collected during the most active 30 minutes of the subject's day between the final randomized treatment phase measurement (mean of endpoint data collected each day during week 8) and baseline phase (mean of endpoint data collected each day during week -1), as measured by wrist-worn accelerometer collected actigraphy (total counts per 30 min period collected during the most active 30 minutes of each day). A ratio > 1 indicates an increase in mean activity counts from baseline to week 8.
Time Frame: Baseline, week 8
Population: Full Analysis Set
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Enalapril | Sacubitril/Valsartan
Number analyzed (Participants) | 60 | 64
Ratio | 1.0411 [0.9938 to 1.0906] | 0.9844 [0.9411 to 1.0297]
Statistical Analysis 1: Comparison: Enalapril vs Sacubitril/Valsartan; Test type: Superiority; p = 0.0895, ANCOVA; model for a log-scaled response with treatment group as a class variable and the baseline value in logarithmic scale as a continuous covariate; Ratio of Geometric Means (SacVal/Ena) = 0.9456, 95% CI 2-sided [0.8863 to 1.0088]

2. Secondary Outcome: Change in Mean Activity Counts During Most Active 30 Minutes of Day From Baseline to Week 1
Description: Change in mean activity counts during most active 30 minutes of day from baseline phase (mean of data collected during week -1) to week 1 (mean of data collected during week 1), as measured by actigraphy (total counts per 30 min period collected during the most active 30 minutes of each day).
Time Frame: Baseline, Week 1
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: counts
Arm/Group | Enalapril | Sacubitril/Valsartan
Number analyzed (Participants) | 54 | 59
counts | 171.3 (440.9) | 464.9 (421.8)
Statistical Analysis 1: Comparison: Enalapril vs Sacubitril/Valsartan; Test type: Superiority; p = 0.6316, ANCOVA; model with treatment group as a class variable and the baseline value as a continuous covariate; Mean Difference (Net) = 293.6, 95% CI 2-sided [-916.5 to 1503.8]

3. Secondary Outcome: Change in Mean Activity Counts During Most Active 30 Minutes of Day From Baseline to Week 9 and 16
Description: Change in mean activity counts during most active 30 minutes of day from baseline phase (mean of data collected during week -1 for Sacubitril/Valsartan and mean of data collected during week 8 for Enalapril) to week 9 and 16 (mean of data collected during weeks 9 and 16), as measured by actigraphy (total counts per 30 min period collected during the most active 30 minutes of each day).
Time Frame: Baseline (Sacubitril/Valsartan: week -1/ Enalapril: week 8), week 9 and 16
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: counts
Arm/Group | Enalapril | Sacubitril/Valsartan
Number analyzed (Participants) | 62 | 64
counts
  Week 9 (change from Baseline): number analyzed (Participants) | 54 | 58
  Week 9 (change from Baseline) | -198.8 (5245.5) | -402.9 (5857.0)
  Week 16 (change from Baseline): number analyzed (Participants) | 51 | 55
  Week 16 (change from Baseline) | -455.1 (4966.7) | 46.9 (4811.2)

4. Secondary Outcome: Change in Mean Activity (Counts Per Minute) During Sleep From Baseline to Week 8
Description: Change in mean activity (counts per minute) during sleep from baseline phase (mean of data collected during week -1) to the final randomized treatment phase measurement (mean of data collected during week 8), as measured by actigraphy (activity counts per minute during daily sleep period, wrist-worn accelerometer).
Time Frame: Baseline, Week 8
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: counts/minute
Arm/Group | Enalapril | Sacubitril/Valsartan
Number analyzed (Participants) | 64 | 65
counts/minute | 0.339 (0.752) | 2.377 (0.746)
Statistical Analysis 1: Comparison: Enalapril vs Sacubitril/Valsartan; Test type: Superiority; p = 0.0570, ANCOVA; model with treatment group as a class variable and the baseline value as a continuous covariate; Mean Difference (Net) = 2.038, 95% CI 2-sided [-0.062 to 4.138]

5. Secondary Outcome: Change in Mean Activity (Counts Per Minute) During Sleep From Baseline to Week 1
Description: Change in mean activity (counts per minute) during sleep from baseline phase (mean of data collected during week -1) to week 1 (mean of data collected during week 1), as measured by actigraphy (activity counts per minute during daily sleep period, wrist-worn accelerometer).
Time Frame: Baseline, Week 1
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: counts/minute
Arm/Group | Enalapril | Sacubitril/Valsartan
Number analyzed (Participants) | 59 | 63
counts/minute | 0.169 (0.696) | 2.647 (0.674)
Statistical Analysis 1: Comparison: Enalapril vs Sacubitril/Valsartan; Test type: Superiority; p = 0.0121, ANCOVA; model with treatment group as a class variable and the baseline value as a continuous covariate; Mean Difference (Net) = 2.478, 95% CI 2-sided [0.553 to 4.403]

6. Secondary Outcome: Change in Mean Activity (Counts Per Minute) During Sleep From Baseline to Week 9 and 16
Description: Change in mean activity (counts per minute) during sleep from baseline phase (mean of data collected during week -1 for Sacubitril/Valsartan and mean of data collected during week 8 for Enalapril) to week 9 and 16 (mean of data collected during week 9 and 16), as measured by actigraphy (activity counts per minute during daily sleep period, wrist-worn accelerometer).
Time Frame: Baseline (Sacubitril/Valsartan: week -1 / Enalapril: week 8), week 9 and 16
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: counts/minute
Arm/Group | Enalapril | Sacubitril/Valsartan
Number analyzed (Participants) | 62 | 64
counts/minute
  Week 9 (change from Baseline): number analyzed (Participants) | 52 | 56
  Week 9 (change from Baseline) | 2.158 (5.150) | 3.230 (7.269)
  Week 16 (change from Baseline): number analyzed (Participants) | 56 | 60
  Week 16 (change from Baseline) | 1.066 (5.367) | 1.489 (5.642)

ADVERSE EVENTS:
Time Frame: 8 weeks in Randomized Treatment Period (Week 1 - Week 8). 8 Weeks in Open-Label Extension Period (Week 9 - Week 16)
Groups:
- Enalapril (Randomized Treatment Period): Week 1 to Week 8: Enalapril
- Sacubitril/Valsartan (Randomized Treatment Period): Week 1 to Week 8: Sacubitril/Valsartan
- Enalapril (Open-Label Extension Period); Sacubitril/Valsartan (Open-Label Extension Period): Week 9 - 16: Sacubitril/Valsartan
Arm/Group | Enalapril (Randomized Treatment Period) | Sacubitril/Valsartan (Randomized Treatment Period) | Enalapril (Open-Label Extension Period) | Sacubitril/Valsartan (Open-Label Extension Period)
All-Cause Mortality (participants affected / at risk) | 1/70 | 0/69 | 0/62 | 0/64
Serious Adverse Events (participants affected / at risk) | 4/70 | 5/69 | 4/62 | 3/64
Other Adverse Events (participants affected / at risk) | 26/70 | 8/69 | 11/62 | 11/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Enalapril (Randomized Treatment Period) (N=70) | Sacubitril/Valsartan (Randomized Treatment Period) (N=69) | Enalapril (Open-Label Extension Period) (N=62) | Sacubitril/Valsartan (Open-Label Extension Period) (N=64)
Angina pectoris (Cardiac disorders) | 1 | 1 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 1 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 1 | 0 | 0 | 0
Complication associated with device (General disorders) | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0 | 0
Incoherent (Nervous system disorders) | 0 | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1 | 0 | 1
Peripheral coldness (Vascular disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Enalapril (Randomized Treatment Period) (N=70) | Sacubitril/Valsartan (Randomized Treatment Period) (N=69) | Enalapril (Open-Label Extension Period) (N=62) | Sacubitril/Valsartan (Open-Label Extension Period) (N=64)
Diarrhoea (Gastrointestinal disorders) | 6 | 1 | 2 | 1
Vomiting (Gastrointestinal disorders) | 4 | 0 | 1 | 0
Fatigue (General disorders) | 9 | 1 | 1 | 5
Dizziness (Nervous system disorders) | 12 | 5 | 5 | 4
Hypotension (Vascular disorders) | 4 | 1 | 4 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-03-13): https://cdn.clinicaltrials.gov/large-docs/69/NCT02970669/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-10): https://cdn.clinicaltrials.gov/large-docs/69/NCT02970669/SAP_001.pdf